CLINICAL TRIAL: NCT05138432
Title: More Fresh Fruit and Vegetable Prescription Program for Families With Type 2 Diabetes Mellitus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency); Rady Children's Hospital, San Diego (Other)
Responsible Party: Principal Investigator, Kay Rhee, Professor of Pediatrics, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1027421
Record Dates: First submitted 2021-11-08; First posted 2021-12-01 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Fruit

STUDY DESIGN:
Intervention Model Description: Participants upon enrollment will be randomized into two groups, either to immediately receive up to $105 per month in vouchers for 12 months (intervention group) or to receive $105 per month in incentives for 12 months after a 6-month delay (delayed-intervention group)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Other): Monthly fruit and vegetable vouchers for 12 months, to start immediately after enrollment.
  Interventions: Behavioral: Fruit and Vegetable Prescription Voucher
- Delayed Intervention Group (Other): Monthly fruit and vegetable vouchers for 12 months, to start after a 6-month waiting period.
  Interventions: Behavioral: Fruit and Vegetable Prescription Voucher

INTERVENTIONS:
Behavioral: Fruit and Vegetable Prescription Voucher — Each participant will immediately (intervention group) or after a 6-month waiting period (delayed-intervention group) receive seven $15 vouchers (value $105 per month) for 12 months. Up to 4 vouchers ($60 total) can be redeemed at any one transaction for purchase of fresh fruits and vegetables, dried beans and legumes at participating Northgate Gonzalez markets. Both groups will continue to receive diabetes and nutrition education as is standard in their practice.

SUMMARY:
Rady Children's Hospital San Diego (RCHSD), UCSD Division of Child and Community Health and the Center for Community Health, and Northgate Gonzalez (NG) Markets will collaborate to create a Produce Prescription Program (Fruit and Vegetable Prescription Program) to be implemented in the RCHSD Diabetes Clinic. We will provide families on Medi-Cal who have a child with T2DM with a fruit and vegetable prescription (FVRx) which will enhance their ability to purchase GusNIP-eligible fresh fruits and vegetables (FV). These prescriptions will be delivered in the form of an electronic voucher that can be filled at any NG Markets throughout San Diego and Riverside counties. The goal of this program is to increase the purchase and consumption of fresh fruits and vegetables, decrease food insecurity, and improve metabolic outcomes for children with type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
Participants upon enrollment will be randomized into two groups, either to immediately receive nutrition incentive vouchers for 12 months (intervention group) or to receive nutrition incentive vouchers for 12 months after a 6-month delay (delayed-intervention group). To evaluate the implementation and outcomes of this program, we will collect fruit and vegetable prescription (FVRx) voucher data in addition to standardized laboratory studies, (hemoglobin A1c (HbA1c), total cholesterol, HDL cholesterol and liver function tests (LFTs)) and physiologic assessments (height, weight) at the child's follow-up appointments through the Diabetes Clinic. These markers will be evaluated at baseline, 6-, 12- and 18-months. Additionally, we will ask participants to complete online or phone surveys including the Dietary Screener Questionnaire (DSQ) for youth and parents and the 18-item US Household Food Security Survey Module every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age < 18 years old
* Diagnosis of type 2 diabetes mellitus
* Hemoglobin A1c greater than or equal to 6.5
* Receiving care at the Rady Children's Hospital Diabetes Clinic

Exclusion Criteria:

* Another immediate family member living in the same household who is already recruited into the study

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Household food security | Survey will be completed at baseline and 12 months
  18-item US Household Food Security Survey Module
Change in Hemoglobin A1c | Measured as part of the participant's routine care in the Diabetes Clinic at baseline and 12 months
  Point of care A1c

SECONDARY OUTCOMES:
Change in BMI z-score | Measured at baseline and 12 months as part of the participant's routine care in the Diabetes Clinic
  BMI calculated by measured height and weight and converted to BMI z-score
Change in Total cholesterol | Measured at baseline and 12 months as part of the participant's routine care in the Diabetes Clinic
  Serum Total cholesterol
Change in Liver function tests | Measured at baseline and 12 months as part of the participant's routine care in the Diabetes Clinic
  Serum aspartate transaminase (AST), serum alanine transaminase (ALT)
Change in Blood pressure | Measured at baseline and 12 months as part of the participant's routine care in the Diabetes Clinic
  Systolic and diastolic BP
Change in beta carotene | Measured at baseline and 12 months
  serum beta carotene levels
Change in fruit and vegetable intake | Survey will be completed at baseline and 12 months.
  Change in child fruit and vegetable intake as measured by the DSQ
Change in HDL cholesterol | Measured at baseline and 12 months as part of the participant's routine care in the Diabetes Clinic
  Serum HDL cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Rhee, MD, MS, MA, Principal Investigator — University of California San Diego, Rady Children's Hospital San Diego
Locations (1):
- Rady Children's Hospital San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No